CLINICAL TRIAL: NCT03443102
Title: The 15-year Impact of Severe Acute Respiratory Syndrome on Organ Functions, Exercise Capacity, and Quality of Life in Survivors.
Brief Title: Long-term Assessment of Organ Functions Among Survivors of Severe Acute Respiratory Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhancheng Gao, Head of Respiartory and Critical Care Medicine, Peking University People's Hospital
Other Study IDs: 2018PHB010-01
Record Dates: First submitted 2018-02-04; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: SARS Virus; Long-Term Survivors
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells would be extracted from participators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS survivors: First-line HCWs infected during the SRAS-CoV pandemic in Peking University People's Hospital, China. Diagnose was further confirmed by SARS-CoV seropositive results.
- Controls: 1. Coworkers of the infected HCWs, who also exposed to SARS patients or specimens. Infection was further excluded by SARS-CoV seronegative results.
  2. Healthy controls matched for age, sex and disease condition, but without exposures to SARS virus.

SUMMARY:
SARS-CoV has caused severe epidemic respiratory disease in human populations. By July 2003, a total of 8,096 probable cases of SARS had been reported including 774 deaths in 27 countries, around one-third of which were health care workers (HCWs). Previous studies have been reported about long-term impacts of SARS infection, including lung function deficiency, steroid-induced osteonecrosis, reduced exercise capacity, and impairment in health-related quality of life (HRQoL). HCWs, especially nurses, have been reported to experience greater psychological distress, particularly increased levels of posttraumatic stress symptomatology (PTSS). But the very complex impacts of this fatal infection on HCWs have not been fully elucidated. It is thus important to follow these occupational patients to detect and manage multi-organ sequelae and functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers who were working at Peking University People's Hospital during the SARS epidemic in 2002-2003

Exclusion Criteria:

* Refusal to continue the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care workers who were working at Peking University People's Hospital during the SARS epidemic in 2002-2003 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause disability | Evaluations would be finished within 90 days after enrollment.
  Disabilities arising from physical injuries and/or mental stresses

SECONDARY OUTCOMES:
Cardiopulmonary function | Evaluations would be finished within 90 days after enrollment.
  The interrelationship between the workings of the heart and lung organs would be assessed by assessed by 6MWT (6-min walk test)
Life Life quaities mental distress | Evaluations would be finished within 90 days after enrollment.
  Quality of life would be assessed by the Medical Outcomes Study 36-item short form version 2 (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Baoguo Jiang, Dr, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li J, Zheng Y, Zhao L, Yue Z, Pan F, Chen Y, Yu B, Chen Y, Zhao G, Zhou Y, Gao Z. Investigation of the impact of SARS-CoV infection on the immunologic status and lung function after 15 years. BMC Infect Dis. 2021 Nov 24;21(1):1183. doi: 10.1186/s12879-021-06881-3. PMID 34819019